CLINICAL TRIAL: NCT01211925
Title: Distal Venous Arterialisation in the Treatment of Critical Ischemia of Lower Limb
Brief Title: Distal Venous Arterialisation of Ischemic Limb
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Clinic for Vascular and Endovascular Surgery, Clinical Center of Serbia, Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 440/III-3
Record Dates: First submitted 2010-09-16; First posted 2010-09-30 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Critical Limb Ischemia
Keywords: unreconstructable peripheral arterial disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- critical ischemia (Experimental)
  Interventions: Procedure: distal venous arterialisation
- Control (No Intervention): Best medical treatment
  Interventions: Drug: Aspirin

INTERVENTIONS:
Procedure: distal venous arterialisation — The investigators perform reverse revascularisation of the ischemic limb with arterial blood supply from patent in flow artery to the superficial dorsal venous arch.
  Other Names: Venous arterialisation, arteriovenous reversal
  Arms: critical ischemia
Drug: Aspirin — 100 mg per day continuous
  Arms: Control

SUMMARY:
Distal venous arterialisation (DVA) improve outcome in patients with nonreconstructible peripheral arterial occlusive disease.

DETAILED DESCRIPTION:
The aim of this study was to estimate validity of distal venous arterialisation (DVA) as a limb salvage procedure. This prospective randomized study reported early results of 30 unreconstructible patients with critical limb ischemia (CLI) treated during 2009 year at Clinic for vascular surgery, Clinical Center of Serbia in Belgrade. Patients were divided in two groups, 10 treated with DVA and 20 conservatively (CT) using antiplatelet drugs.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any possibility for direct revascularisation due to extensive occlusive disease of crural and pedal arteries
* Sufficient deep venous system and usable great saphenous vein as a graft for in situ bypass surgery according duplex scanning
* localized infective of necrotic process up to the metatarsal level
* Satisfactory general patient condition

Exclusion Criteria:

* advanced lower limb ischemia
* venous insufficiency of lower limb

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
limb salvage | 1 year
  The investigators will estimate clinical improvement in patients with critical limb ischemia underwent of distal venous arterialisation. Comparative group consist patients treated with antiplatelet drugs.

SECONDARY OUTCOMES:
lactate level in the blood of deep venous system | 1 year
  The investigators measure metabolic changes in the patients after distal venous arterialisation

CONTACTS AND LOCATIONS:
Overall Officials: Predrag Vl Djoric, MD, Principal Investigator — Clinical Center of Serbia in Belgrade, Clinic for Vascular and Endovascular Surgery
Locations (1):
- Clinical Center of Serbia, Belgrade, Serbia, Serbia